CLINICAL TRIAL: NCT02766777
Title: A Multicenter, 6-month, Open-label Safety Study of Lubiprostone in Pediatric Subjects Aged ≥ 6 Years to < 18 Years With Functional Constipation
Brief Title: Evaluation of the Safety of Lubiprostone in Pediatric Participants Aged ≥ 6 Years to < 18 Years With Functional Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo AG (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCMP-0211-303
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lubiprostone (Experimental): Participants received lubiprostone twice daily (BID). Participants received either lubiprostone 12 mcg BID, lubiprostone 24 mcg BID (dose based on participant's weight) up to 24 weeks.
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 12 or 24 mcg soft capsules for oral administration.
  Other Names: Amitiza

SUMMARY:
A study of the safety of lubiprostone in pediatric participants aged ≥ 6 Years to < 18 years diagnosed with functional constipation.

DETAILED DESCRIPTION:
To assess the long-term safety and tolerability of oral lubiprostone 12 or 24mcg capsules dosed twice daily (BID) when administered orally for 24 weeks in pediatric participants with functional constipation. Evaluation of lubiprostone safety and tolerability is the primary objective in this study.

ELIGIBILITY:
Inclusion Criteria:

* Medically-confirmed diagnosis of Functional Constipation per Rome III Diagnostic Criteria for Childhood Functional Constipation
* At least 6 years of age but less than 18 years of age at the time of randomisation
* Only stable dose of selective serotonin re-uptake inhibitors (SSRIs), serotonin-specific reuptake inhibitor (SNRIs), or monoamine oxidase inhibitors (MAO) inhibitors are allowed if participant is taking antidepressants

Exclusion Criteria:

* Any gastrointestinal (GI) condition, other than constipation, affecting GI motility or defecation
* Untreated faecal impaction at the time of screening
* Medical/surgical condition that might interfere with the absorption, distribution, metabolism, or excretion of the study medication

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (13):
- United States (13):
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - Methodist Medical Center, Peoria, Illinois
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - Pioneer Clinical Research, Bellevue, Nebraska
  - PriMed Clinical Research, Beavercreek, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Coastal Clinical Research, Charleston, South Carolina
  - Coastal Pediatrics Associates - Mount Pleasant, Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - 3rd Coast Research Associates, Corpus Christi, Texas
  - Bridgerland Clinical Research, Logan, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lubiprostone
Started | 87
Treated (Safety [SAF] Population) | 87
Completed | 53
Not Completed | 34
Not completed — Adverse Event | 12
Not completed — Lost to Follow-up | 16
Not completed — Non-Compliance With Study Drug | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Safety (SAF) population, defined as all enrolled participants who took at least one dose of study medication.
Arm/Group | Lubiprostone
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (3.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 16
  White | 68
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: Adverse events with onset dates after the administration of the first dose of study medication or prior to the last day of treatment plus 7 days are considered treatment-emergent.
Time Frame: within 25 weeks
Population: Safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Lubiprostone: Participants received lubiprostone 12 mcg or 24 mcg BID (dose based on participant's weight) up to 24 weeks.
Arm/Group | Lubiprostone
Number analyzed (Participants) | 87
Participants | 47

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 25 weeks
Arm/Group | Lubiprostone
All-Cause Mortality (participants affected / at risk) | 0/87
Serious Adverse Events (participants affected / at risk) | 2/87
Other Adverse Events (participants affected / at risk) | 24/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=87)
Colitis ulcerative (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=87)
Diarrhoea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Blood iron decreased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes